CLINICAL TRIAL: NCT01393678
Title: A Multicenter, Randomized, Double-blind, 2 Parallel Group, Phase 3 Study of PENNEL Capsule in Chronic Liver Disease
Brief Title: Study to Evaluate Efficacy and Safety of PENNEL Capsule in the Patients With Chronic Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: R&D department, CR team
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMK-PENNEL 3
Record Dates: First submitted 2011-07-03; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PENNEL (Experimental): 2cap T.I.D
  Interventions: Drug: PENNEL
- NISSEL (Active Comparator): NISSEL
  BDD (biphenylmethyl dicarboxylate) ................25mg
  2cap T.I.D
  Interventions: Drug: NISSEL

INTERVENTIONS:
Drug: NISSEL — Biphenyl Dimethyl Dicarboxylate 25mg ............. 1 cap
  Arms: NISSEL
Drug: PENNEL — Biphenyl Dimethyl Dicarboxylate 25mg & garlic oil 50mg ............. 1cap
  Arms: PENNEL

SUMMARY:
The drug in this study is combined product of biphenyl dimethyl dicarboxylate (DDB) and garlic oil. This components showed synergistic enhancing effects in previous tests. In phase 2 test, 6 cap three times a day dosage (2cap T.I.D) is better than other dosage. Based on above, this study is phase 3 test to prove efficacy and safety of PENNEL.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic hepatitis by biopsy
* Patients over 20, under 65 years of age.
* Patients with abnormal transaminase value.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients who have any history of esophageal bleeding, hepatic encephalopathy, ascites.
* Diabetes, thyroid dysfunction, fatty liver, liver cancer patients.
* Toxic hepatitis, alcoholic hepatitis.
* Total bilirubin value more than 3.0 mg/dl.
* Albumin value less than 3.0 g/dl.
* Patients who participating in other study about drug.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 1997-11; Primary Completion 1998-03 (Actual); Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
ALT(Alanine Aminotransferase) | 10 weeks
  To evaluate the efficacy of the PENNEL capsule on change ALT from baseline to 10 weeks (Change from Baseline in Alanine Aminotransferase at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration

SECONDARY OUTCOMES:
AST (Aspartate Aminotransferase) | 10 weeks
  To evaluate the efficacy of the PENNEL capsule on change AST from baseline to 10 weeks(Change from Baseline in Aspartate Aminotransferase at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration
g-GT (γ-glutamyl transpeptidase) | 10 weeks
  To evaluate the efficacy of the PENNEL capsule on change g-GT from baseline to 10 weeks (Change from Baseline in γ-glutamyl transpeptidase at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration
Total bilirubin | 10 weeks
  To evaluate the efficacy of the PENNEL capsule on change Total bilirubin from baseline to 10 weeks (Change from Baseline in Total bilirubin at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration
PLT (Platelet) | 10 weeks
  To evaluate the efficacy of the PENNEL capsule on change PLT from baseline to 10 weeks (Change from Baseline in Platelet count at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration
Total cholesterol | 10 weeks
  To evaluate the efficacy of the Oltipraz on change Total cholesterol from baseline to 10 weeks (Change from Baseline in Total cholesterol at 10 weeks)
  The measurements were conducted four times, including ① before administration, ② the 4th week of administration, ③ the 8th week of administration ④ the 10th week of administration

CONTACTS AND LOCATIONS:
Overall Officials: Minho Lee, MD.PhD, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Hospital, Seoul, Seongdong-gu,, South Korea